CLINICAL TRIAL: NCT03864848
Title: ENRAPT-MR Trial: Epicardial Mitral Repair
Brief Title: Epicardial Mitral Repair Trial - ENRAPT-MR
Acronym: ENRAPT-MR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mitre Medical Corp. (Industry)
Collaborators: Meditrial Europe Ltd. (Industry); Medical Metrics Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPL-0001
Record Dates: First submitted 2018-11-01; First posted 2019-03-06 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Intervention Model Description: Registry
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Treatment (Experimental): Treatment with the Mitral Touch Implant for Epicardial Annuloplasty.
  Interventions: Device: Mitral Touch Implant

INTERVENTIONS:
Device: Mitral Touch Implant — The study population for this study will be comprised of patients who are to undergo cardiac surgery with a sternotomy (e.g. CABG) and who present moderate to severe ischemic or functional MR. In order to be considered eligible for the study, each patient must meet the conditions listed in the inclusion and none of the exclusion criteria.

SUMMARY:
Mitral Touch System

This device is designed to epicardially reshape the mitral valve annulus without the need for cardiopulmonary bypass (CPB) and open heart access (atriotomy), in patients with left ventricular dilation and ischemic or functional MR (mitral regurgitation (MR)).

DETAILED DESCRIPTION:
Mitre Medical has developed an epicardial mitral annuloplasty device that can be implanted concomitant during planned coronary artery bypass surgery to help treat the MR patients. The Mitral Touch is designed to restore the S-L dimension and has the advantage of being placed without stopping the heart and placing the patient on a bypass pump.

ELIGIBILITY:
Inclusion Criteria:

* Patient has moderate (2+), moderate-to-severe (3+) or severe (4+) ischemic or functional Mitral regurgitation per 2D or 3D echocardiography, symptomatic or asymptomatic
* Patient is 18 years of age or older
* Patient is willing and able to sign informed consent form

Exclusion Criteria:

* History of endocarditis or current endocarditis
* Structural abnormalities of the leaflets and papillary muscles*
* Dysfunctional chordae*
* Any prior cardiac surgery including but not limited to CABG, Mitral Valve repair surgery, mechanical prosthetic Valve, or ventricular assist device, prior sternotomy*
* Ejection fraction <25%
* New York Hheart Association (NYHA) class IV
* MV diameters > 7cm
* Myxomatous Mitral regurgitation
* Renal insufficiency (eGFR < 30 ml/min)
* Severely calcified (posterior) Mitral Valve annulus
* Women who are pregnant (by history of menstrual period or pregnancy test if history is considered unreliable)
* Any coronary artery calcification at site of placement as determined by angiogram.
* Abnormal cardiac anatomy discovered prior to surgery or during procedure.
* Pericardial adhesions

  * NOTE: Patients with prior or concurrent mitral chordae repair (example: PTFE or Neochord) are potential candidates for the MitralTouch

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-12-18 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Safety - 30 - Day Major Adverse Event Rate | 30-Days
  30 - Day Major Adverse Event Rate All-cause mortality Stroke Life-threatening bleeding (MVARC scale) Major vascular complications Major cardiac structural complications Stage 2 or 3 acute kidney injury (includes new dialysis) Severe hypotension, worsening of heart failure, or respiratory failure requiring intravenous pressors or invasive or mechanical heart failure treatments such as ultrafiltration or hemodynamic assist devices, including intra-aortic balloon pumps or left ventricular or biventricular assist devices, or prolonged intubation for >48 h Emergency surgery or re-intervention related to the device or access procedure

SECONDARY OUTCOMES:
Technical Success - MR Reduction | 30-Days, 6 Months, 12 Months
  MR assessment of MR Grade by TTE compared to baseline
Technical Success - Coaptation Length Increase | 30-Days, 6 Months, 12 Months
  An increase of coaptation length compared to baseline
Technical Success - Septa-Lateral Reduction | Implantation, 6 Months, 12 Months
  Target of 15%-30% Reduction when compared to baseline
Technical Success - Improvement in NYHA Classification | 6 & 12 Months
  Reduction in NYHA Classification compared to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Vilnius University Hospital Santariskiu Klinikos, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Takaseya T, Shiose A, Saraiva RM, Fumoto H, Arakawa Y, Juravic M, Lombardi P, Fukamachi K. Novel epicardial off-pump device for mitral regurgitation: acute evaluation. Eur J Cardiothorac Surg. 2010 Jun;37(6):1291-6. doi: 10.1016/j.ejcts.2009.11.054. PMID 20137971
- [Background] Takaseya T, Fumoto H, Saraiva RM, Shiose A, Arakawa Y, Park M, Rao S, Dessoffy R, Kramer LD Jr, Juravic M, Lombardi P, Fukamachi K. Acute feasibility study of a novel device for the treatment of mitral regurgitation in a normal canine model. Innovations (Phila). 2010 Jan;5(1):28-32. doi: 10.1097/IMI.0b013e3181cdf735. PMID 22437273
- [Result] Thourani VH, George I, Rucinskas K, Kalinauskas G, Janusauskas V, Zakarkaite D, Ailawadi G, Smith R, Mack MJ. First in human experience with an epicardial beating heart device for secondary mitral regurgitation. J Thorac Cardiovasc Surg. 2021 Mar;161(3):949-958.e4. doi: 10.1016/j.jtcvs.2020.11.169. Epub 2020 Dec 14. PMID 33436291